CLINICAL TRIAL: NCT02301065
Title: Analysis of KIR+CD56+ T Cells and FcRg-CD56+CD3- NK Cells in Pediatric Allogeneic Hematopoietic Stem Cell Transplant Patients and Donors
Brief Title: Analysis of T Cell and Natural Killer (NK) Cell in Relation to Viral Infections in Pediatric Stem Cell Transplant Patients and Donors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Sponsor
Other Study IDs: KIRT
Record Dates: First submitted 2014-11-18; First posted 2014-11-25 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Hematologic Malignancies
Keywords: Viral; Infection; Allogeneic Stem Cell Transplant
MeSH Terms: conditions — Hematologic Neoplasms; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stem Cell Donors: Allogeneic hematopoietic stem cell transplant (HSCT) donors. Blood samples for phenotypes research will be collected once from donors, prior to apheresis for collection of donor stem cells.
- Stem Cell Recipients: Allogeneic hematopoietic stem cell transplant (HSCT) recipients. Blood samples will be drawn prior to transplantation and every two weeks, up to day 100 post-transplantation.

SUMMARY:
Viral infections and reactivation during pediatric allogeneic hematopoietic stem cell transplantation (HSCT) are a common occurrence and significantly contribute to post-transplant morbidity and mortality. The risk is high due to prolonged periods of immune deficiency while awaiting immune reconstitution post-transplant. Current strategies to reduce complications from viral infections include prophylactic treatment, close monitoring for viral infections and prompt treatment at the first sign of symptoms or increasing viral load. However, the most definitive treatment for viral infections remains the host's cellular defenses. Improved understanding of the immune systems response to viral infections may lead to better treatment strategies.

This study is being done to explore the relationships between T-cells and NK cells (infection fighting cells) and viral infections or reactivations in young allogeneic stem cell transplant patients. The investigators will be looking at how these cells react and function in young patients receiving allogeneic stem cell transplantation, as well as in healthy stem cell donors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* To explore the expansion patterns of KIR+CD56+ T-cells and FcRg-CD56+CD3- NK cells in response to viral infection and reactivation in pediatric allogeneic hematopoietic stem cell transplant (HSCT) patients.

SECONDARY OBJECTIVES:

* To describe the phenotype of KIR+CD56+ T-cells and FcRg-CD56+CD3- NK cells in pediatric allogeneic HSCT patients and healthy donors.
* To describe the specificity and functional capacity of KIR+CD56+ T-cells against viral antigens in both pediatric allogeneic HSCT patients and healthy donors.
* To describe the functional capacity of FcRg-CD56+CD3- NK cells against CMV-infected cells in both pediatric allogeneic HSCT patients and healthy donors.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing allogeneic hematopoietic stem cell transplant (HSCT) for a hematologic malignancy or a donor for a patient undergoing allogeneic hematopoietic stem cell transplant for a hematologic malignancy.
* For HSCT patients: ages birth to 21 years old; for donors: any age.
* For minors less than 18 years old, both parents must be available on St. Jude campus to provide consent. One parent/legal guardian will be acceptable if one parent is deceased, incompetent, or when the one parent present has legal responsibility for the care and custody of the child.

Exclusion Criteria:

* Patients undergoing allogeneic hematopoietic stem cell transplant for a disease other than a hematologic malignancy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study is planned to enroll 50 pediatric allogeneic hematopoietic stem cell transplant (HSCT) patients and 50 donors. All patients/donors who meet eligibility criteria and sign the consent form will be enrolled on the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Percentage of KIR+CD45+ T-cells in stem cell recipients and donors | Donors once within 1 week prior to stem cell donation. HSCT recipients: baseline within 1 week prior to stem cell infusion and every 2 weeks, up to 100 days post-transplantation
  Blood samples will be drawn as follows:
  * Donors will have a blood sample drawn once within 1 week prior to stem cell donation.
  * HSCT recipients will have serial blood samples: a baseline sample within 1 week prior to stem cell infusion and collections every 2 weeks, up to 100 days post-transplantation
  Summary statistics of the two cell populations, such as mean, median, range, and standard error, will be provided.
Number of FcRg-CD56+CD3- NK cells in stem cell recipients and donors | Donors once within 1 week prior to stem cell donation. HSCT recipients: baseline within 1 week prior to stem cell infusion and every 2 weeks, up to 100 days post-transplantation
  Blood samples will be drawn as follows:
  * Donors will have a blood sample drawn once within 1 week prior to stem cell donation.
  * HSCT recipients will have serial blood samples: a baseline sample within 1 week prior to stem cell infusion and collections every 2 weeks, up to 100 days post-transplantation
  Summary statistics of the two cell populations, such as mean, median, range, and standard error, will be provided.

SECONDARY OUTCOMES:
Surface marker expression density of phenotype KIR+CD56+ T-cells and FcRg-CD56+CD3- NK cells in donors and recipients | Donors once within 1 week prior to stem cell donation. HSCT recipients: within 1 week prior to stem cell infusion and within 1 week of 100 days post-transplantation
  Blood samples will be drawn as follows:
  * Donors will have a blood sample drawn once within 1 week prior to stem cell donation.
  * HSCT recipients will have two blood samples drawn: the first within 1 week prior to stem cell infusion, and the second within 1 week of 100 days post-transplantation
  Surface marker expression density will be calculated and summary statistics will be provided for all calculations.
Percentage of KIR+CD56+ T-cells that stain for tetramer/pentamer | Donors once within 1 week prior to stem cell donation. HSCT recipients: baseline within 1 week prior to stem cell infusion and every 28 days, up to 100 days post-transplantation
  Blood samples will be drawn as follows:
  * Donors will have percentages measured once within 1 week prior to stem cell donation.
  * HSCT recipients will have serial blood samples, a baseline sample within 1 week prior to stem cell infusion, and collections every 28 days, up to 100 days post-transplantation
  The specificity of KIR+CD56+T-cells will be evaluated through viral tetramer/pentamer staining.
Change in numbers and percentages of KIR+CD56+T-cells after exposure to viral antigen in vitro and cytokine expression levels | Donors once within 1 week prior to stem cell donation. HSCT recipients: baseline within 1 week prior to stem cell infusion and every 28 days, up to 100 days post-transplantation
  Blood samples will be drawn as follows:
  * Donors will have a blood sample drawn once within 1 week prior to stem cell donation.
  * HSCT recipients will have serial blood samples, including a baseline sample within 1 week prior to stem cell infusion and collections every 28 days, up to 100 days post-transplantation
  The functional capacity of KIR+CD56+T-cells will be evaluated through proliferation and cytokine production assays. Summary statistics will be provided.
Number of FcRg-CD56+CD3- NK cells after exposure to cytomegalovirus | Donors once within 1 week prior to stem cell donation. HSCT recipients: within 1 week prior to stem cell infusion and within 1 week of 100 days post-transplantation
  Blood samples will be drawn as follows:
  * Donors will have will have one blood sample drawn within 1 week prior to stem cell donation.
  * HSCT recipients will have two blood samples drawn: the first within 1 week prior to stem cell infusion, and the second within 1 week of 100 days post-transplantation
  Summary statistics of the functional capacity of FcRg-CD56+CD3- NK against CMV-infected cells will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Talleur, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols